CLINICAL TRIAL: NCT01419314
Title: Lower Extremity Splinting to Manage Pain and Sleep Disturbances Associated With HIV/AIDS Related Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Harris County Hospital District (Other Government); DJO Incorporated (Industry)
Responsible Party: Principal Investigator, Robert Sandoval, Principal Investigator, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16196
Record Dates: First submitted 2011-08-10; First posted 2011-08-18 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: HIV; AIDS; Peripheral Neuropathy; Pain; Sleep
Keywords: Physical Therapy; Splint; Sleep; Pain; 6 min walk; forward reach; Function
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Splinting application (Experimental): Participants will be asked to wear a pair of LE night splints for the duration of the study (6 weeks) at night/during sleep only.
  Interventions: Device: Splinting application to the lower extremities
- Splint liner application (Placebo Comparator): The liner or protective sheath from the Walkabout™ splint will be applied to the LEs, with the structural frame of the splint removed by the researcher in advance, patients will be blinded to this arm of the study.
  Interventions: Device: Splint liner application

INTERVENTIONS:
Device: Splinting application to the lower extremities — Walkabout™ splints (Don Joy Orthopedics, Vista, CA, USA) will used in the splinting treatment. The Walkabout splint is a one-piece injection molded walking boot fitted with a rocker bottom allowing for ambulation. The participants will be fitted and instructed to wear the bilateral LE splints to sleep for the duration of the study (6 weeks).
  Other Names: Walkabout splint
  Arms: Splinting application
Device: Splint liner application — The liner or protective sheath from the Walkabout™ splint will be applied to the LEs, with the structural frame of the splint removed by the researcher in advance, patients will be blinded to this arm of the study (6 weeks).
  Other Names: Walkabout liner
  Arms: Splint liner application

SUMMARY:
WHAT IS THE PURPOSE OF THIS STUDY? The investigators want to know if wearing a pair of splints at night works to bring the pain down and help you sleep better (in people living with HIV/AIDS related neuropathy).

HOW MANY PEOPLE WILL PARTICIPATE? About 58 to 88 people will take part in this study at the Harris County Hospital District (HCHD).

WHAT WILL HAPPEN DURING THIS STUDY? As a participant, you will be assigned to one of two treatment groups. In one group, you will be asked to wear leg splints at night and the other you will wear the liners of the splints only.

You will be asked to answer questions about how well you sleep, how long you sleep, and about your discomfort at the legs. The researcher will be there to help, but the investigators want you to answer the questions on your own if you can. You will be asked to reach forwards standing next to a wall and to walk for 6 minutes after that. The tests will de done in random order. The sessions will be done at the beginning, at week three and week six. You should finish all of the testing and questionnaires in an hour or less, for a total of three hours over six weeks in the investigators clinic.

You will receive instructions on how to use the splints with liners or the liners alone at home. You will be asked to wear them at night only for the next 6 weeks. Finally, the principal investigator will contact you weekly by phone, to discuss issues of comfort and your ability to adhere to the instructions provided.

DETAILED DESCRIPTION:
The medical management of people living with the Human Immunodeficiency Virus that ultimately leads to the development of Acquired Immunodeficiency Syndrome has progressed dramatically since the beginning of the pandemic in the early 1980's. Despite advances in management and prevention, it is estimated that 33 million people worldwide are infected with this virus. Of those, 1.1 million people living with HIV/AIDS reside in the United States, while 56,000 new cases are added to this total every year. Medical providers are challenged to achieve a delicate balance between offering effective anti-retroviral therapeutic interventions while monitoring undesired side effects in an aging population of "People Living with HIV/AIDS" (PLWA). Indeed, the life expectancy of PLWA has continued to increase in the industrialized world, approaching parity with non-infected individuals.

Pain and sleep disturbances are commonly associated with chronic systemic diseases such as fibromyalgia, arthritis, chronic liver disease and HIV/AIDS. Data collected from a cohort of 317 PLWA, indicate that 55% of them experienced and ranked increases in pain and sleep disturbances among the top four symptoms associated with living with HIV/AIDS. Pain and sleep disturbances were only preceded in reported prevalence by self-reported fatigue and drowsiness. A review of systemic diseases' impact on sleep, suggests that alterations in rapid eye movement (REM), non-REM sleep stages, as well as an increase in sleep disturbances are associated with HIV disease progression into AIDS; moreover, 26% of the variance in sleep disturbances experienced by PLWA in that study was attributed to pain and other psychosocial factors.

Peripheral neuropathy (PN) is among the most common complications associated with long-term survival with HIV/AIDS. It is estimated that 30-60% of all PLWA will develop PN at some point during the course of the disease, with an increased prevalence seen in this patient population as the disease progresses from HIV into AIDS. Functional impairments have also been reported in the presence of neuropathies. Different authors have reported significant differences in gait quality, walking speed and total distance walked in individuals with damage to the peripheral nervous system. Despite advances in medical management of HIV infection, the direct impact of commonly experienced symptoms associated with living with HIV/AIDS, such as pain and sleep disturbances in the current era of anti-retroviral therapy has not been extensively reported in the literature.

In a recent pilot study, conducted by this author and colleagues, the use of night time lower extremity (LE) splinting showed promising results in the management of pain and sleep disturbances. This pilot study design was a crossover study that included 22 PLWA with PN and evaluated the effects of a three-week bilateral lower splints application on pain and sleep. A 20% improvement in both pain and sleep scores was reported in this pilot study. Additionally, a moderate effect size for pain and sleep scores was found. The results suggested that the analgesic effect of the splint application persisted for a period of several weeks following discontinuation of the lower splint application. These results were obtained using a relatively small sample of patients and without a long-term follow-up post-splinting application. Finally, that study could not determine whether the source of the pain inhibition was due to the application of a full contact protective sheath on the lower leg or the short-term immobilization at the ankle joints provided by the splints.

Purpose and Hypotheses

Therefore, the purpose and primary aim of this study is to evaluate the management of pain and sleep disturbances in people living with HIV/AIDS-related PN with the use of bilateral LE splints versus a control/placebo intervention of bilateral LE splint liner application. The null hypotheses for the primary aim are:

* There is no difference in pain and sleep scores between the bilateral LE splints and those obtained using the splint liners only following a three and six-week application.
* There is no difference in pain and sleep scores between baseline and following a six-week LE splint application.

The secondary aim is to identify factors influencing function, as measured by the functional reach test and the six-minute walk test; and their relationship with pain and sleep disturbances in the presence of HIV/AIDS related neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Adult PLWA 18 and older, with a clinical diagnosis of symptomatic bilateral LE PN will be invited to participate.
* The participants will be on a stable pain and HIV/AIDS management regimen without foreseeable alterations or changes to said pharmacological regimen, which may include pain and or sleep medications.
* The participants will be community dwelling individuals, able to walk at or above a modified independence level with or without the need of an assistive device to ambulate, such as a cane or walker.
* Eligible participants will report at least one of the following clinical symptoms: paresthesia, dysesthesia, and report night cramps in the LE

Exclusion Criteria:

* Participants will be excluded if they have a clinical diagnosis of any of the following: significant cardiovascular or pulmonary disease (specifically, myocardial infarction within the past six months, angina, or dyspnea at rest), paraplegia, hemiplegia, other major neurological dysfunction, diabetes, absent pedal pulse during examination, sleep apnea, or are pregnant.
* Additionally, patients unable to read English, patients with changes to their pharmacological management during the study and or using any mechanical devices to assist in normalizing sleep will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sandoval, MS, PT, Principal Investigator — Texas Woman's University
Locations (1):
- Thomas Street Health Center-HCHD, Houston, Texas, United States

REFERENCES:
- [Background] Sandoval R, Runft B, Roddey T. Pilot study: does lower extremity night splinting assist in the management of painful peripheral neuropathy in the HIV/AIDS population? J Int Assoc Physicians AIDS Care (Chic). 2010 Nov-Dec;9(6):368-81. doi: 10.1177/1545109710373828. Epub 2010 Nov 12. PMID 21075912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were randomized to use a night application of bilateral lower extremity splints (23 participants) or using the soft liners of the splints only (23 participants). One participant was excluded from the liner group as he failed to disclose a recent diabetes diagnosis.
Pre-assignment Details: One of the participants in the liner group was excluded from the study at the beginning as he developed type-II diabetes. The total number of participants in the liner group was thus 22 at baseline.
Groups:
- Splint Liner Application: The liner or protective sheath from the Walkabout™ splint will be applied to the LEs, with the structural frame of the splint removed by the researcher in advance.
Period: Start of Study
Arm/Group | Splinting Application | Splint Liner Application
Started | 23 (minor comfort issues were reported within the first 2 weeks of the trial) | 22 (No comfort issues reported.)
Completed | 23 | 22
Not Completed | 0 | 0
Period: Follow-up at Week 3 of the Trial
Arm/Group | Splinting Application | Splint Liner Application
Started | 23 (3 participants discontinued the trial, 3 failed to return for additional follow-ups.) | 22 (one participant failed to return for the 3 week follow-up)
Completed | 17 | 21
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 3 | 0
Period: Follow-up at Week 6 of the Trial
Arm/Group | Splinting Application | Splint Liner Application
Started | 17 | 21 (2 participants did not return for their final follow-up)
Completed | 16 (2 people who missed the first follow-up, returned for the final follow-up at week 6 (n=18).) | 19
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- LE Splints Group: Participants were asked to wear a pair of LE night splints for the duration of the study (6 weeks) at night/during sleep only.
- Splint Liner Application: The liner or protective sheath from the Walkabout™ splint was applied to the LEs, with the structural frame of the splint removed by the researcher in advance.
- Total: Total of all reporting groups
Arm/Group | LE Splints Group | Splint Liner Application | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 50.65 (8.04) | 46.09 (7.71) | 48.42 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 14 | 12 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 9 | 6 | 15
  Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
CD4 [Mean (Standard Deviation); unit: cells/mm3] — The most recent CD4 cell counts were extracted from the medical record.
  cells/mm3 | 586.13 (233.64) | 446.09 (232.54) | 517.67 (241.07)
Log Viral load [Log Mean (Standard Deviation); unit: Log (copies/ml)] — The most recent measured HIV viral load (log viral load) was extracted from the medical record. Measured in viral copies/ml on a logarithmic scale with 1.48 log/ml representing undetectable viral load levels for the viral load test conducted in our site (less than 50 copies/ml)
  Log (copies/ml) | 2.25 (1.08) | 1.96 (0.75) | 2.10 (0.93)
Years living with HIV [Mean (Standard Deviation); unit: years] — The number of years living with HIV was calculated by subtracting the year of diagnosis to the year of sutdy enrollment.
  years | 11.30 (6.01) | 10.32 (7.62) | 10.82 (6.79)
Pain scores [Mean (Standard Deviation); unit: Scores on a 0-100 scale.] — Neuropathic Pain Scale (NPS) score, where a score of "0" equates to "no pain" and "100" is the maximum neuropathic pain score possible. The scale score is computed by totaling all 10 pain sub-scales, each individually scored from 0-10.
  Scores on a 0-100 scale. | 61.35 (20.98) | 60.16 (14.35) | 60.77 (17.85)
Sleep Scores [Mean (Standard Deviation); unit: Scores on a 0-21 scale] — Pittsburgh Sleep Quality Index (PSQI),this is a 0-21 score scale with 21/21 denoting maximum sleep disturbances. The PSQI is scored by adding all seven sub-scales, each with a maximum score of three. A score greater than 5/21 characterizes the individual as a "poor sleeper."
  Scores on a 0-21 scale | 14.13 (3.89) | 15.14 (4.68) | 14.62 (4.28)
Function- Forward reach [Mean (Standard Deviation); unit: Centimeters (cm)] — The average of 3 reaching trials are reported. One participant in the liner group had extreme reaching values (>3 standard deviation from the mean) and was excluded from the report (n=22). Longer distances in this test represent better volitional control of balance in the sagittal plane. Reaching distances >30 cm are considered to be within normal limits.
  Centimeters (cm) | 35.31 (6.45) | 36.88 (8.36) | 36.07 (7.37)
Function-Walking Distance [Mean (Standard Deviation); unit: Meters (m)] — The 6 minute walk distance was collected on all participants. Longer walking distances represent decreased impact on function. Non-HIV cohorts typically are able to walk 400-600m in six-minutes.
  Meters (m) | 246.00 (133.71) | 241.89 (151.46) | 243.99 (141.04)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores at Week 3
Description: A composite pain score was collected using the self-reported Neuropathic Pain Scale (NPS). In this zero to 100 scale, the participant is asked to quantify the different aspects of the pain experience in the presence of neuropathies.
Time Frame: Week 3
Population: The total number of participants returning for the first follow-up at week three with complete data.
Measure: Mean (Standard Deviation); unit: units on a scale 0-100 (0= no pain)
Groups:
- Lower Extremity Splinting Application: nighttime splint application to the lower extremities
- Splint Liner: Night time application of lower extremity splint liner
Arm/Group | Lower Extremity Splinting Application | Splint Liner
Number analyzed (Participants) | 16 | 21
units on a scale 0-100 (0= no pain) | 50.53 (16.48) | 53.76 (15.41)

2. Primary Outcome: Pain Scores
Description: as for outcome 1
Time Frame: Week 6
Population: The total number of participants that completed the 6 week trial in each investigational group
Measure: Mean (Standard Deviation); unit: units on a scale 0-100 (0=no pain)
Groups:
- Splinting Application: Participants were asked to wear a pair of LE night splints for the duration of the study (6 weeks) at night/during sleep only.
Arm/Group | Splinting Application | Splint Liner Application
Number analyzed (Participants) | 18 | 19
units on a scale 0-100 (0=no pain) | 40.22 (18.57) | 49.89 (21.72)
Statistical Analysis 1: Comparison: Splinting Application vs Splint Liner Application; A repeated measure ANOVA was performed to evaluate the contrasts of interest; Test type: Superiority or Other; p = 0.001, ANOVA; Sphericity was not tenable for the factor pain scores, degrees of freedom were corrected using Huynh-Feldt estimates, df (1.71,56.46); Mean Difference (Final Values) = 45.19, 95% CI 2-sided [38.33 to 52.05], Standard Deviation 20.25
Statistical Analysis 2: Comparison: Splinting Application; Null hypothesis: Is there a difference in baseline pain scores compared to those at week 6 in the splinting group?; Test type: Superiority or Other; p < 0.0005, t-test, 2 sided — Bonferroni adjustment for significance<0.013; Mean Difference (Final Values) = 16.09, 95% CI 2-sided [8.80 to 23.39], Standard Error of Mean 3.60 — Paired t-test contrasting pain scores from baseline to week six of the trial-Splint group. The statistical power for the within splint intervention contrast was calculated to be 0.99
Statistical Analysis 3: Comparison: Splinting Application vs Splint Liner Application; Null Hypothesis: There is not difference in pain scores between the liner and splint applications at week three; Test type: Superiority or Other; p = 0.155, t-test, 2 sided — Bonferroni adjustment for significance<0.013; df(35); Mean Difference (Final Values) = -3.23, 95% CI 2-sided [-13.93 to 7.47], Standard Error of Mean 5.27 — The statistical power for the between intervention contrast was calculated to be 0.26
Statistical Analysis 4: Comparison: Splinting Application vs Splint Liner Application; Null Hypothesis: There is no difference in pain scores between the liner and splint applications at week six; Test type: Superiority or Other; p = 0.155, t-test, 2 sided; df(35); Mean Difference (Final Values) = -9.67, 95% CI 2-sided [-23.20 to 3.85], Standard Error of Mean 6.66

3. Secondary Outcome: Function-Reach
Description: Forward reach test
  For this test, the investigators asked the participants to stand next to a wall without shoes and with their feet positioned hip-width apart on the floor with one shoulder close to the wall. The participants were instructed "to reach as far forward as possible, without losing your balance, touching the wall or stepping and crossing the tile threshold on the floor". The average distance of three reaching attempts was recorded and used in the analysis.
Time Frame: week 3
Population: The number of participants returning for the first follow-up. One participant in the liner group had baseline scores greater than 3 standard deviation difference from the mean and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Lower Extremity Splinting Application | Splint Liner
Number analyzed (Participants) | 16 | 20
Centimeters (cm) | 38.76 (6.76) | 38.35 (7.04)

4. Secondary Outcome: Function-Reach
Description: as for outcome 3
Time Frame: week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Lower Extremity Splinting Application | Splint Liner
Number analyzed (Participants) | 18 | 18
Centimeters (cm) | 40.00 (6.22) | 39.34 (6.22)

5. Primary Outcome: Sleep Quality/Quantity Scores (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a ten item questionnaire, covering the following seven components of sleep: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunctions.
Time Frame: week 3
Population: The number of participants returning for the first follow-up with complete data.
Measure: Mean (Standard Deviation); unit: Scores ranging 0-21, 0=no disturbances
Arm/Group | Splinting Application | Splint Liner Application
Number analyzed (Participants) | 16 | 21
Scores ranging 0-21, 0=no disturbances | 13.13 (4.51) | 14.29 (4.58)

6. Primary Outcome: Sleep Quality/Quantity Scores (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a ten item questionnaire, covering the following seven components of sleep: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunctions. Buysse et al. reported sensitivity and specificity values of 89.6% and 86.5%, respectively for this scale in identifying good and poor sleepers.
Time Frame: week 6
Population: The number of participants returning for the second follow-up
Measure: Mean (Standard Deviation); unit: Scores ranging 0-21, 0=no disturbances
Arm/Group | Splinting Application | Splint Liner Application
Number analyzed (Participants) | 18 | 19
Scores ranging 0-21, 0=no disturbances | 12.06 (4.84) | 11.95 (5.57)

7. Secondary Outcome: Function-Walking Distance
Description: Six minute walk test
  For this test the participants were instructed to: "Please walk as far, as fast and as safe as you can for up to six minutes". The walking test will be performed in a climate-controlled environment, on a level surface void of obstacles and with a pre-determined path of 68 feet (or approximately 20 m) per lap. The beginning and end of the 34-foot path were clearly marked with taped trapezoids to the non-skid floor.
Time Frame: week 3
Population: The number of participants returning for the 3 week follow-up with complete data
Measure: Mean (Standard Deviation); unit: Meters (m)
Arm/Group | Lower Extremity Splinting Application | Splint Liner
Number analyzed (Participants) | 16 | 19
Meters (m) | 255.84 (143.58) | 263.52 (156.74)

8. Secondary Outcome: Function-Walking Distance
Description: as for outcome 7
Time Frame: week 6
Population: The number of participants returning for the 6 week follow-up
Measure: Mean (Standard Deviation); unit: Meters (m)
Arm/Group | Lower Extremity Splinting Application | Splint Liner
Number analyzed (Participants) | 18 | 19
Meters (m) | 279.52 (146.61) | 304.90 (137.63)

ADVERSE EVENTS:
Arm/Group | Lower Extremity Splinting Application | Splint Liner
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
The contrast between the splinting group and liner group was statistically underpowered. The data was collected and analyzed by the primary investigator. The clinical diagnosis of peripheral neuropathy was not confirmed with EMG or punch skin biopsy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No